CLINICAL TRIAL: NCT00651482
Title: Treatment of Refractory Metastatic Renal Cell Carcinoma With Bevacizumab and RAD001 (Everolimus)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Sandy Srinivas (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Sandy Srinivas, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-11789; RENAL0016 (Other: OnCore); 98593 (Other: Stanford University Alternate IRB Approval Number); AVF4304s (Other: Genentech-Roche); 41839 (Other: Novartis, Inc)
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Kidney Neoplasms; Kidney (Renal Cell) Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab + RAD001 (everolimus) (Experimental): Study treatment, consisting of bevacizumab + everolimus, was administered as 28-day cycles
  Bevacizumab 10 mg/kg administered by IV infusion every 14 days (dose suspension permitted, dose reduction not permitted)
  Everolimus 10 mg daily was administered orally (dose reduction to 5 mg daily and then 5 mg every other day, was permitted as needed for toxicity or tolerability)
  Interventions: Drug: Everolimus; Drug: Bevacizumab

INTERVENTIONS:
Drug: Everolimus
  Other Names: Zortress; Certican; RAD001
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
To determine the safety and efficacy of the combination of bevacizumab and everolimus (RAD001) for the treatment of metastatic renal cell cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically confirmed metastatic RCC that is predominantly clear cell Measurable disease, as defined by RECIST
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* No more than 1 prior targeted therapy (eg, sorafenib, sunitinib) (prior cytokine therapy allowed)
* No more than 2 prior systemic therapies
* Ability and capacity to comply with the study and follow-up procedures

General Exclusion Criteria

* Inability to comply with study and/or follow-up procedures
* Life expectancy of < 12 weeks
* Inadequate organ function, as evidenced by any of the following at screening:

  * Absolute neutrophil count (ANC) < 1500/uL
  * Platelet count ≤ 100 x 10^9/L
  * Total bilirubin ≥ 1.5 x upper limit of normal (ULN)
  * AST and/or ALT > 2.5 x ULN for patients without evidence of liver metastases, or 5 x ULN for patients with documented liver metastases
  * Serum creatinine > 2.0 mg/dL
  * Hemoglobin < 9 g/dL (may be transfused or receive epoetin alfa to maintain or exceed this level)
* Active infection or fever > 38.5°C within 3 days of starting treatment
* Women who are pregnant or breast feeding,
* Able to conceive and unwilling to practice an effective method of birth control.
* History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, early-stage bladder cancer, or low-grade endometrial cancer
* Malignancies that have undergone a putative surgical cure (i.e., localized prostate cancer post-prostatectomy) within 5 years prior to Day 1 may be discussed with the Principal Investigator.
* Any other medical conditions (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a patient's ability to provide informed consent, cooperate, or participate in the study, or to interfere with the interpretation of the results.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study

Disease-Specific Exclusion Criteria

* RCC with predominantly sarcomatoid features
* Radiotherapy for RCC within 28 days prior to Day 1, with the exception of single-fraction radiotherapy given for the indication of pain control
* Prior treatment with bevacizumab or any mTOR inhibitor (eg, temsirolimus, sirolimus, or everolimus)
* Current need for dialysis

Bevacizumab-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known CNS disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Significant vascular disease (eg, aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy that is not intentionally pharmacologically-induced
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by a urine protein:
* Creatinine (UPC) ratio ≥ 1.0. If UPC ratio ≥ 1.0, the patient must undergo a 24 hour urine collection which must demonstrate ≤ 1g of protein in 24 hours to be eligible.
* Known hypersensitivity to any component of bevacizumab

RAD001-Specific Exclusion Criteria

* Known hypersensitivity to any component of RAD001
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Severely impaired lung function (spirometry and DLCO < 50% of normal and O2 saturation 88% or less at rest on room air)
* If O2 saturation is ≤ 88% at rest on screening, pulmonary function tests (PFTs) will be ordered to confirm normal pulmonary function and eligibility.
* Fasting total cholesterol > 350 mg/dL
* Fasting triglyceride level > 400 mg/dL or >2.5 x ULN
* Fasting serum glucose > 250 mg/dL
* Serum phosphorus < 2.0 mg/dL
* Serum corrected calcium < 8.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Harshman LC, Barbeau S, McMillian A, Srinivas S. A phase II study of bevacizumab and everolimus as treatment for refractory metastatic renal cell carcinoma. Clin Genitourin Cancer. 2013 Jun;11(2):100-6. doi: 10.1016/j.clgc.2012.12.002. Epub 2013 Jan 24. PMID 23352238

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + RAD001 (Everolimus): Study treatment, consisting of bevacizumab + everolimus, was administered as 28-day cycles
  Bevacizumab 10 mg/kg administered by IV infusion every 14 days (dose suspension permitted, dose reduction not permitted)
  Everolimus 10 mg daily was administered orally (dose reduction to 5 mg daily and then 5 mg every other day, was permitted as needed for toxicity or tolerability)
  Everolimus
  Bevacizumab
Period: Overall Study
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 55 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response (OR)
Description: Number of subjects with objective response (OR)
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
participants | 1

2. Secondary Outcome: Objective Response (OR) Duration
Time Frame: 24 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
weeks | 21.7 [13.0 to 50.0]

3. Secondary Outcome: Time-to-Treatment Failure (TTF)
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
months | 5.1 [1.9 to 11.7]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: 44 months
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
months | 21.0 [4.8 to 43.8]

5. Secondary Outcome: Number of Subjects With Drug-related SAEs
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
participants | 3

6. Secondary Outcome: Total Number of Drug-related SAEs
Time Frame: 24 months
Measure: Number; unit: events
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
events | 4

7. Secondary Outcome: Treatment Discontinuation Due to Toxicity
Description: Number of subjects whose treatment was discontinued due to toxicity
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
participants | 4

8. Secondary Outcome: Treatment Discontinuation Due to Disease Progression
Description: Number of subjects whose treatment was discontinued due to disease progression
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
participants | 6

9. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) per RECIST criteria
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Number analyzed (Participants) | 10
months | 5.1 [3.1 to 11.7]

ADVERSE EVENTS:
Arm/Group | Bevacizumab + RAD001 (Everolimus)
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + RAD001 (Everolimus) (N=10)
Blood and lymphatic system disorders - Other, Thrombotic microangiopath (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal disorders - Inferior vena cava obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pain - Resection of left distal femur; ORIF of supracondylar fracture (General disorders) | 1 (1)
Pain - Right hip pain progressively worsened (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Fracture - Avulsion fractue of the lesser trochanter of R femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular disorders - GI hemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + RAD001 (Everolimus) (N=10)
Anemia (Blood and lymphatic system disorders) | 10 (37)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 6 (8)
Hemolysis (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 3 (5)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (27)
Nausea (Gastrointestinal disorders) | 5 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 3 (4)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 9 (13)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6)
Alkaline phosphatase increased (Investigations) | 6 (12)
Aspartate aminotransferase increased (Investigations) | 6 (14)
Blood bilirubin increased (Investigations) | 1 (2)
Cholesterol high (Investigations) | 5 (15)
CPK increased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 9 (17)
INR increased (Investigations) | 1 (2)
Investigations - Other (Investigations) | 4 (6)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 4 (8)
Weight gain (Investigations) | 1 (3)
Weight loss (Investigations) | 5 (7)
White blood cell decreased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (20)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 (18)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (27)
Hypokalemia (Metabolism and nutrition disorders) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 7 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (5)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Sinus pain (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Chronic kidney disease (Renal and urinary disorders) | 3 (4)
Hematuria (Renal and urinary disorders) | 8 (15)
Proteinuria (Renal and urinary disorders) | 10 (37)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (9)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No